CLINICAL TRIAL: NCT00140582
Title: Advanced Follicular Lymphoma Evaluating the Benefit of Maintenance Therapy With Rituximab (MabThera®) After Induction of Response With Chemotherapy Plus Rituximab in Comparison With no Maintenance Therapy
Brief Title: Primary Rituximab and Maintenance
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Lymphoma Study Association (Other)
Collaborators: HOVON - Dutch Haemato-Oncology Association (Other); German Low Grade Lymphoma Study Group (Other); Australasian Leukaemia and Lymphoma Group (Other); Institute of Cancer Research, United Kingdom (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRIMA
Record Dates: First submitted 2005-08-22; First posted 2005-09-01 (Estimated); Last update posted 2017-03-13 (Actual); Status verified 2017-03

CONDITIONS: Follicular Lymphoma
Keywords: lymphoma; follicular; maintenance
MeSH Terms: conditions — Lymphoma, Follicular; Lymphoma | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A : rituximab maintenance (Experimental): Maintenance with rituximab for 2 years
  Interventions: Drug: Rituximab
- B : no maintenance (No Intervention): No further treatment

INTERVENTIONS:
Drug: Rituximab — rituximab 375 mg/m2 every 8 weeks for 24 months (12 injections) or control with no treatment
  Arms: A : rituximab maintenance

SUMMARY:
* Objectives

  * Primary objective: To evaluate in patients with advanced follicular lymphoma the benefit of maintenance therapy with rituximab after induction of response with chemotherapy plus rituximab in comparison with no maintenance therapy
  * Secondary objective: To evaluate response rates, event driven survival endpoints (EFS, PFS, OS) and quality of life of four different chemotherapy regimens combined with rituximab, with or without maintenance with rituximab, for first line treatment of advanced stage follicular lymphoma.
* Study Design This is an international open-label, multicentre, randomized study with two treatment phases. In the induction phase patients have to respond to 1st line induction treatment in order to be eligible for randomization to the second phase of maintenance treatment or observation. After the maintenance period patients will be included in the follow up phase for 3 years.

DETAILED DESCRIPTION:
Study medication

* First period: Induction of response with 8 x rituximab combined with 8 cycles of CVP or 6 cycles of CHOP in 21-day cycles or 6 cycles of FCM in 28-day cycles or 6 cycles of MCP in 28-day cycles.
* Second period: rituximab 375 mg/m2 every 8 weeks for 24 months (12 injections) or control with no treatment

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed follicular lymphoma grade 1, 2 or 3a.
* Patients previously untreated.
* Patients with at least one of the following symptoms requiring initiation of treatment:

  * Bulky disease at study entry according to the GELF criteria: nodal or extranodal mass > 7cm in its greater diameter
  * B symptoms
  * Elevated serum LDH or beta2-microglobulin
  * involvement of at least 3 nodal sites (each with a diameter greater than 3 cm)
  * symptomatic splenic enlargement
  * compressive syndrome
  * pleural/peritoneal effusion
* Age must be > 18 years.
* Performance status < 2 on the ECOG scale (see appendix E).
* Adequate hematological function within 28 days prior to registration (unless those abnormalities are related to lymphoma extension), this includes:

  * Hemoglobin ≥ 8.0 g/dl (5.0 mmol/L)
  * Absolute neutrophil count (ANC) ≥ 1.5 109/L
  * Platelet count ≥ 100 109/L
* Women are not breast feeding, are using effective contraception, are not pregnant and agree not to become pregnant during participation in the trial and during the 12 months thereafter. Men agree not to father a child during participation in the trial and during the 12 months thereafter.
* Having previously signed a written informed consent form.

Exclusion Criteria:

* Transformation to high-grade lymphoma (secondary to "low-grade" follicular lymphoma).
* Grade 3b follicular lymphoma.
* Presence or history of CNS disease (either CNS lymphoma or lymphomatous meningitis).
* Patients regularly taking corticosteroids during the last 4 weeks, unless administered at a dose equivalent to < 20 mg/day prednisone.
* Patients with prior or concomitant malignancies except non-melanoma skin cancer or adequately treated in situ cervical cancer.
* Major surgery (excluding lymph node biopsy) within 28 days prior to registration.
* Poor renal function: Serum creatinine > 2.0 mg/dl (197 μmol/L),
* Poor hepatic function: total bilirubin > 2.0 mg/dl (34 μmol/L), AST (SGOT) > 3 x the upper limit of normal unless these abnormalities are related to lymphoma.
* Known HIV infection or active HBV or HCV infection.
* Serious underlying medical conditions, which could impair the ability of the patient to participate in the trial (e.g. ongoing infection, uncontrolled diabetes mellitus, gastric ulcers, active autoimmune disease). Judgment is up to the investigator.
* Life expectancy < 6 months
* Known sensitivity or allergy to murine products
* Treatment within a clinical trial within 30 days prior to trial entry
* Adult patient under tutelage.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1217 (Actual)
Dates: Start 2004-12 (Actual); Primary Completion 2007-05 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | number of event observed driven : 344 events or 10 years
  defined as the time from randomization to progression, relapse, death from any cause.

SECONDARY OUTCOMES:
Response rates, event driven survival endpoints (EFS, PFS, OS) | number of event observed driven : 344 events or 10 years
Quality of life | number of event observed driven : 344 events or 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Gilles A Salles, MD PhD, Principal Investigator — Lymphoma Study Association
Locations (24):
- Fundaleu Hospital, Buenos Aires, Argentina
- Australian Leukemia and Lymphoma Group, Melbourne, Australia
- Belgium (2):
  - Université de Gent, Ghent
  - Groupe d'Etude des Lymphomes de l'adulte, Mont-Godinne
- Hospital Samaritano, São Paulo, Brazil
- Fundación Santafé de Bogotá, Bogotá, Colombia
- Amtssygehuset i Herlev, Herlev, Denmark
- France (12):
  - Polyclinique Bordeaux Nord, Bordeaux
  - Hôpital Henri Mondor, Créteil
  - Hématologie CHU de Lille, Lille
  - Centre Léon Bérard, Lyon
  - Institut Curie, Paris
  - Hôpital Saint Louis, Paris
  - Hématologie Adultes - Hôpital Necker, Paris
  - Service d'Hématologie - Centre Hospitalier Lyon-Sud, Pierre-Bénite
  - Centre Hospitalier Robert Debré, Reims
  - Centre Henri Becquerel, Rouen
  - Hématologie CHU Purpan, Toulouse
  - Institut Gustave Roussy, Villejuif
- HOVON, Utrecht, Netherlands
- Australia New Zealand Leukemia Lymphoma Group, Auckland, New Zealand
- Instituo Nacional de Enfermedades Neoplasicas, Lima, Peru
- Hospital Clinic Barcelona, Barcelona, Spain
- King Chulalongkorn Memorial Hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bachy E, Seymour JF, Feugier P, Offner F, Lopez-Guillermo A, Belada D, Xerri L, Catalano JV, Brice P, Lemonnier F, Martin A, Casasnovas O, Pedersen LM, Dorvaux V, Simpson D, Leppa S, Gabarre J, da Silva MG, Glaisner S, Ysebaert L, Vekhoff A, Intragumtornchai T, Le Gouill S, Lister A, Estell JA, Milone G, Sonet A, Farhi J, Zeuner H, Tilly H, Salles G. Sustained Progression-Free Survival Benefit of Rituximab Maintenance in Patients With Follicular Lymphoma: Long-Term Results of the PRIMA Study. J Clin Oncol. 2019 Nov 1;37(31):2815-2824. doi: 10.1200/JCO.19.01073. Epub 2019 Jul 24. PMID 31339826
- [Derived] Zhou X, Wang J, Zhang J, Copley-Merriman C, Torigoe Y, Reyes C, Seymour JF, Offner FC, Trneny M, Salles GA. Symptoms and toxicity of rituximab maintenance relative to observation following immunochemotherapy in patients with follicular lymphoma. Hematology. 2015 Apr;20(3):129-36. doi: 10.1179/1607845414Y.0000000179. Epub 2014 Jul 16. PMID 25029908
- [Derived] Ghesquieres H, Cartron G, Seymour JF, Delfau-Larue MH, Offner F, Soubeyran P, Perrot A, Brice P, Bouabdallah R, Sonet A, Dupuis J, Casasnovas O, Catalano JV, Delmer A, Jardin F, Verney A, Dartigues P, Salles G. Clinical outcome of patients with follicular lymphoma receiving chemoimmunotherapy in the PRIMA study is not affected by FCGR3A and FCGR2A polymorphisms. Blood. 2012 Sep 27;120(13):2650-7. doi: 10.1182/blood-2012-05-431825. Epub 2012 Aug 10. PMID 22885164
- [Derived] Salles G, Seymour JF, Offner F, Lopez-Guillermo A, Belada D, Xerri L, Feugier P, Bouabdallah R, Catalano JV, Brice P, Caballero D, Haioun C, Pedersen LM, Delmer A, Simpson D, Leppa S, Soubeyran P, Hagenbeek A, Casasnovas O, Intragumtornchai T, Ferme C, da Silva MG, Sebban C, Lister A, Estell JA, Milone G, Sonet A, Mendila M, Coiffier B, Tilly H. Rituximab maintenance for 2 years in patients with high tumour burden follicular lymphoma responding to rituximab plus chemotherapy (PRIMA): a phase 3, randomised controlled trial. Lancet. 2011 Jan 1;377(9759):42-51. doi: 10.1016/S0140-6736(10)62175-7. Epub 2010 Dec 20. PMID 21176949
- See also: Related Info — http://www.gela.org